CLINICAL TRIAL: NCT03728244
Title: Clinical Comparison of MEBO Ointment and Hyaluronic Acid Gel in the Management of Pain After Free Gingival Graft Harvesting: A Randomized Clinical Trial
Brief Title: MEBO Ointment and Hyaluronic Acid Gel in the Management of Pain After Free Gingival Graft Harvesting
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Hassan, postgraduate student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170992
Record Dates: First submitted 2018-10-27; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Graft Pain; Gingival Recession
Keywords: mucoginival defects; Free gingival graft; palatal donor site; pain
MeSH Terms: conditions — Gingival Recession; Pain | interventions — gamma-sitosterol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- test group Hyaluronic acid (Experimental): Patients scheduled for free gingival graft harvesting will receive Hyaluronic acid gel 0.2%
  Interventions: Drug: Hyaluronic Acid gel
- test group MEBO ointment (Experimental): Patients scheduled for free gingival graft harvesting will receive MEBO ointment
  Interventions: Drug: MEBO ointment
- negative control group (No Intervention): Patients scheduled for free gingival graft harvesting

INTERVENTIONS:
Drug: MEBO ointment — The pharmacological effects of MEBO are attributable to beta-sitosterol, isolated from phellodendron amurense, flavonoids mainly baicalin isolated from scutellaria baicalensis, alkaloids mainly berberine, isolated from coptis chinensi, Beeswax and sesame oil (Zhang et al., 2005).
  Other Names: beta-sitosterol
  Arms: test group MEBO ointment
Drug: Hyaluronic Acid gel — Hyaluronic acid is a substance that is naturally present in the human body. It is found in the highest concentrations in fluids in the eyes and joints. The hyaluronic acid that is used as medicine is extracted from rooster combs or made by bacteria in the laboratory.
  Other Names: gengigel
  Arms: test group Hyaluronic acid

SUMMARY:
Postoperative pain as well as bleeding are the most common complications after palatal graft harvesting also postsurgical swelling have been reported , Although different agents were used to protect the denuded areas on the palate as gelatin sponge , platelet rich fibrin (PRF) , medicinal plant extract (MPE) and platelet concentrate , no gold standard can be specified for this purpose

PICO Format:

P: Patients with mucogingival defects that require free gingival graft. I:1. Hyaluronic acid gel 0.2% placed in the palatal donor site then covered with periodontal pack (test group I) 2.MEBO ointment placed in the palatal donor site then covered with periodontal pack (test group II) C: Periodontal pack only O: Post-operative pain T: day 3, 7, 14, 21 and 42 postoperative.

Aim of the study:

To compare the effect of MEBO ointment versus Hyaluronic acid gel 0.2% applied to palatal donor site in post-operative pain reduction after free gingival graft harvesting.

Research question:

Is MEBO ointment as effective as hyaluronic acid gel in the management of postoperative pain after free gingival graft harvesting in the management of mucogingival defects?

DETAILED DESCRIPTION:
Interventions:

1. Hyaluronic acid gel 0.2%
2. MEBO ointment

Procedure:

The palatal sites will be anaesthetized with 0.3 ml of a solution of 4% Articaine and 0.001% Adrenalin. Graft harvesting will be performed by basic surgical techniques previously described by Miller (1982). A rectangular shaped piece of mucosa will be harvested from the area of the hard palate by a split-thickness dissection.

The graft will then be used as it on the recipient bed.

The graft dimensions will be recorded (width and length).

Denuded palatal area will then be protected using one of the following options:

1. Periodontal pack only (control group)
2. HA gel 0.2% covered with a periodontal pack (test group I)
3. MEBO ointment covered with a periodontal pack (test group II)

Postoperative instructions:

Postoperative instructions will include discontinuing toothbrushing and flossing around the surgical sites until the day of periodontal dressing removal (day 7).

Patients will be directed to consume only soft foods during the first week and to avoid any mechanical trauma.

Patients will be scheduled to be seen on days 3, 7, 14, 21 and 42.

Periodontal pack will be first removed on day 3, and donor sites will be evaluated using selected parameters in both groups.

After evaluation, HA gels together with periodontal pack will be reapplied in test group I, MEBO ointment with periodontal pack will be reapplied in test group II whereas periodontal pack only will be reapplied in control group

On day 7, the periodontal packs will be removed for reevaluation of the wound area in all groups. Thereafter, all patients will be followed up on days 14, 21 and 42 for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mucogingival defects scheduled for free gingival graft
* Systemically healthy

Exclusion Criteria:

* Smokers
* Occlusal trauma at site of graft
* Pregnancy and lactation
* Patients allergic to the used agents
* Severe gagging reflex

Ages: 21 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Post operative pain: VAS | on day 7
  measured by Visual analogue scale between 0 and 10. (0: no pain, 1: minimal pain, 5:moderate pain, 10: severe pain )

SECONDARY OUTCOMES:
Color match | On day 42
  of the palatal mucosa will be assessed by comparing it with that of the adjacent and opposite side by using the objective VAS (VAS score 0-10) represented by a continuous line, by a clinician blinded to the treatment group assignment.
wound size | at day 21
  To be recorded using (UNC 15) periodontal probe to the nearest measurement of 0.5 mm , length and width only

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ang ES, Lee ST, Gan CS, See P, Chan YH, Ng LH, Machin D. The role of alternative therapy in the management of partial thickness burns of the face--experience with the use of moist exposed burn ointment (MEBO) compared with silver sulphadiazine. Ann Acad Med Singap. 2000 Jan;29(1):7-10. PMID 10748957
- [Background] Farnoush A. Techniques for the protection and coverage of the donor sites in free soft tissue grafts. J Periodontol. 1978 Aug;49(8):403-5. doi: 10.1902/jop.1978.49.8.403. PMID 288907
- [Background] Fawzy El-Sayed KM, Dahaba MA, Aboul-Ela S, Darhous MS. Local application of hyaluronan gel in conjunction with periodontal surgery: a randomized controlled trial. Clin Oral Investig. 2012 Aug;16(4):1229-36. doi: 10.1007/s00784-011-0630-z. Epub 2011 Oct 20. PMID 22012469
- [Background] Hammad HM, Hammad MM, Abdelhadi IN, Khalifeh MS. Effects of topically applied agents on intra-oral wound healing in a rat model: a clinical and histomorphometric study. Int J Dent Hyg. 2011 Feb;9(1):9-16. doi: 10.1111/j.1601-5037.2009.00410.x. PMID 21226845
- [Background] Hirsch T, Ashkar W, Schumacher O, Steinstraesser L, Ingianni G, Cedidi CC. Moist Exposed Burn Ointment (MEBO) in partial thickness burns - a randomized, comparative open mono-center study on the efficacy of dermaheal (MEBO) ointment on thermal 2nd degree burns compared to conventional therapy. Eur J Med Res. 2008 Nov 24;13(11):505-10. PMID 19073386
- [Background] Keceli HG, Aylikci BU, Koseoglu S, Dolgun A. Evaluation of palatal donor site haemostasis and wound healing after free gingival graft surgery. J Clin Periodontol. 2015 Jun;42(6):582-9. doi: 10.1111/jcpe.12404. Epub 2015 May 19. PMID 25892528
- [Background] Madi M, Kassem A. Topical simvastatin gel as a novel therapeutic modality for palatal donor site wound healing following free gingival graft procedure. Acta Odontol Scand. 2018 Apr;76(3):212-219. doi: 10.1080/00016357.2017.1403648. Epub 2017 Nov 16. PMID 29145771
- [Background] Patel PV, Kumar S, Vidya GD, Patel A, Holmes JC, Kumar V. Cytological assessment of healing palatal donor site wounds and grafted gingival wounds after application of ozonated oil: an eighteen-month randomized controlled clinical trial. Acta Cytol. 2012;56(3):277-84. doi: 10.1159/000336889. Epub 2012 Apr 26. PMID 22555530
- [Background] Yildirim S, Ozener HO, Dogan B, Kuru B. Effect of topically applied hyaluronic acid on pain and palatal epithelial wound healing: An examiner-masked, randomized, controlled clinical trial. J Periodontol. 2018 Jan;89(1):36-45. doi: 10.1902/jop.2017.170105. PMID 28914592